CLINICAL TRIAL: NCT02780258
Title: Restylane Silk for Photoaged Thinned Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skin Laser & Surgery Specialists (Other)
Responsible Party: Principal Investigator, David J. Goldberg, MD, David J. Goldberg, MD, JD, Skin Laser & Surgery Specialists
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RESTHANDS01
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Photoaged Thinning of the Hands

ARMS (2):
- Restylane Silk Treated Hand (Experimental): The dorsal aspect of one hand will be injected with Restylane Silk.
  Interventions: Device: Restylane Silk
- Control Hand (No Intervention): The dorsal aspect of the hand that is not treated will be used for baseline comparison.

INTERVENTIONS:
Device: Restylane Silk
  Arms: Restylane Silk Treated Hand

SUMMARY:
To evaluate the safety and efficacy of Restylane Silk for photoaged thinned hands

ELIGIBILITY:
Inclusion Criteria:

* Female volunteer
* Aged from 40-70 years on the day of screening
* No known medical conditions that may interfere with study participation
* Moderate to very severe Photoaged thinning of the hands based on the 5-point hand grading scale
* Willingness to not use any products on their hands for the duration of the study
* Read, understand, and sign informed consent forms
* Willingness to sign photography release form
* Willing and able to comply with all follow-up requirements
* Willingness to undergo Restylane Silk injections to one hand

Exclusion Criteria:

* Any significant skin disease at treatment area
* Any medical condition which could interfere with the treatment
* Inability or unwillingness to follow the treatment schedule
* Inability or unwillingness to sign the informed consent
* History of poor wound healing
* History of keloid formation
* History of HIV, hepatitis, immuno-compromised
* Pregnant or lactating
* Previous use of deep chemical peels on the treatment area
* Previous injections of Restylane Silk to the hands
* Known hypersensitivity to Restylane Silk or any of its ingredients
* Previous laser or light based treatments to the treatment area 6 months prior to the screening visit

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Change in photoaged thinning of the treatment area as measured by the 5 point hand grading scale | Baseline, 1month, 3months, 6 months